CLINICAL TRIAL: NCT03642652
Title: Repeated Automated Mobile Text Reminders for Follow-up of Positive Fecal Occult Blood Tests: a Randomized Controlled Trial
Brief Title: SMS Reminders for Positive FOBT Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meuhedet. Healthcare Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 01-023-03-16
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomisation into Intervention and control groups. Text message sent to Intervention group. No intervention in control group
Who Masked: Participant, Care Provider
Masking Description: Participants were not aware of the trial. Only Intervention arm participants received text reminders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS (Experimental): Each patient in the intervention group also received an automated text message up to a week after the positive FOBT result. The text read: "Hello. There is a lab test result ready for you. Contact your physician for an explanation of the findings." Two additional automated text message reminders were sent to the patient at 2 weeks and 1 month reading, "Hello, This is a reminder. It is essential that you contact your physician if you have not already done so."
  Interventions: Behavioral: SMS
- Control (No Intervention): Routine care

INTERVENTIONS:
Behavioral: SMS — Text reminders to mobile telephone
  Other Names: mobile text reminder
  Arms: SMS

SUMMARY:
A randomized controlled trial to examine the effect of 3 mobile telephone text message reminders on followup colonoscopy 120 days after a positive fecal occult blood test among Meuhedet members aged 50-74 who tested positive in 2016.

DETAILED DESCRIPTION:
Background: Fecal occult blood tests are recommended by the US Preventive Services Task Force as a screening method for colorectal cancer, but they are only effective if positive results are followed by colonoscopy. Surprisingly, a large proportion of patients with a positive result do not follow this recommendation.

Objective: To examine the effectiveness of a short message service in increasing adherence to colonoscopy follow-up after a positive fecal occult blood test.

Methods: This randomized controlled trial was conducted with patients who had positive colorectal cancer screening results. Randomization was stratified by residential district and socioeconomic status. Subjects in the control group (n = 238) received routine care that included an alert to the physician regarding the positive Fecal occult blood test result. The intervention group (n = 232) received routine care and three short message service reminders to visit their primary care physician. Adherence to colonoscopy was measured 120 days from the positive result. All patient information, including test results and colonoscopy completion, were obtained from their computerized medical records. Physicians of the study patients completed an attitude survey regarding FOBT as a screening test for colorectal cancer. The intervention and control groups were compared using chi-squared for discrete variables. Logistic regression was used to calculate odds ratios and 95% confidence intervals for performing colonoscopy within 120 days, adjusting for potential confounders of age, gender, socioeconomic status, district, ethnicity, intervention group and physician's attitude.

ELIGIBILITY:
Inclusion Criteria:

* positive fecal occult blood test (FOBT) in 2016
* agreed to receive SMS from healthcare provider

Exclusion Criteria:

* Existing oncology diagnosis
* personal or family history of colorectal cancer
* colonoscopy up to 10 years prior to FOBT

Ages: 50 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Follow-up colonoscopy 120 days after a positive fecal occult blood test | 120 days after positive FOBT
  Completion of colonoscopy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azulay R, Valinsky L, Hershkowitz F, Magnezi R. Repeated Automated Mobile Text Messaging Reminders for Follow-Up of Positive Fecal Occult Blood Tests: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 5;7(2):e11114. doi: 10.2196/11114. PMID 30720439